CLINICAL TRIAL: NCT01871896
Title: Apollo OverStitch for Bariatric Surgery Revision After Weight Loss Failure
Brief Title: Endoscopic Surgery for Bariatric Revision After Weight Loss Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EndoSurgery
Record Dates: First submitted 2013-05-11; First posted 2013-06-07 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Morbid Obesity; Weight Loss
Keywords: Surgical Endoscopy; Morbid Obesity; Weight Loss; Bariatrics; Surgical Revision
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight Gain (Experimental): Patients who previously underwent bariatric surgery who failed to lose the expected weight or regained weight.
  Interventions: Device: Endoscopic Suturing to Create Early Satiety

INTERVENTIONS:
Device: Endoscopic Suturing to Create Early Satiety — Evaluating the efficacy of endoscopic suturing for weight loss.
  Other Names: Endoscopic Cerclage; Bariatric Surgery Revision; Apollo EndoStitch; Apollo OverTube

SUMMARY:
Morbid obesity and its associated metabolic diseases are on the rise in the United States. Currently, the best treatment for obesity is bariatric surgery where both roux-en-Y gastric bypass and sleeve gastrectomy offer substantial weight loss. Unfortunately, 20% of patients who undergo bariatric surgery fail to lose enough weight defined as less than 50% of excess body weight loss or regain of weight. For those patients who fail to lose weight after bariatric surgery and have failed maximal medical therapy and diet supervision, the treatment is re-operation and revision. Re-operation of the abdomen carries significant postoperative morbidity and mortality. The investigators propose to use the Apollo OverStitch endoscopic suturing device that has already been approved by the FDA as an option for bariatric surgery revision without having to re-operate on the patient. The investigators believe that the endoscopic technique may be able to provide weight loss without having to re-operate on the patient.

DETAILED DESCRIPTION:
The most effective weight loss procedures in the United States are both roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (SG)where the majority are performed laparoscopically. Estimated excess body weight loss (EBWL) is >50% at the end of one year. However, nearly 20% of patients fail to meet the estimated EBWL or they may experience weight gain recidivism. The first step is nutritional counseling, medically supervised diets, and medical therapy. Surgery would be for those who still fail to lose weight despite the aforementioned efforts.

It is hypothesized that failure of weight loss for RYGB is gastrojejunostomy (GJ) dilation defined as >2 cm. Surgical treatment would require revision of this dilation. Unfortunately many of these revision procedures cannot be done laparoscopically given dense intra-abdominal adhesions. This will require conversion to an open surgery in a morbidly obese patient thus raising postoperative morbidity and mortality estimated to range between 15%-50%.

The investigators propose to use the endoscopic suturing device designed by Apollo EndoSurgery to decrease the GJ dilation to 5-6 mm thus causing restriction, delayed food transit time, and promote early satiety. These efforts will limit overall caloric intake thereby promoting weight loss.

It is thought that patients with previous SG may have a dilation of their stomach. The investigators propose a pyloric cerclage using the Apollo EndoSurgery suturing device by decreasing the opening of the pylorus thus achieving the same goals that the investigators proposed above with RYGB revision.

Endoscopic procedures are same day procedures with little morbidity and mortality when compared to laparoscopic or open bariatric surgery revision.

ELIGIBILITY:
Inclusion Criteria:

* Previous Roux-En-Y Gastric Bypass (RYGB) or Sleeve Gastrectomy (SG)
* Failure to lose >50% of their excess body weight after 1 year
* Failure of weight loss despite maximal medical therapy and medically-supervised diets

Exclusion Criteria:

* Esophageal Stricture
* Marginal Ulcer at the gastrojejunostomy anastomosis
* Non-compliance with bariatric follow-up
* Gastric ulcers
* Paraesophageal hernias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Rogers, MD, Principal Investigator — University of California, San Francisco; Jonathan T Carter, MD, Principal Investigator — University of California, San Francisco; John P Cello, MD, Principal Investigator — University of California, San Francisco; Matthew Lin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Thompson CC, Chand B, Chen YK, DeMarco DC, Miller L, Schweitzer M, Rothstein RI, Lautz DB, Slattery J, Ryan MB, Brethauer S, Schauer P, Mitchell MC, Starpoli A, Haber GB, Catalano MF, Edmundowicz S, Fagnant AM, Kaplan LM, Roslin MS. Endoscopic suturing for transoral outlet reduction increases weight loss after Roux-en-Y gastric bypass surgery. Gastroenterology. 2013 Jul;145(1):129-137.e3. doi: 10.1053/j.gastro.2013.04.002. Epub 2013 Apr 5. PMID 23567348
- [Background] Deylgat B, D'Hondt M, Pottel H, Vansteenkiste F, Van Rooy F, Devriendt D. Indications, safety, and feasibility of conversion of failed bariatric surgery to Roux-en-Y gastric bypass: a retrospective comparative study with primary laparoscopic Roux-en-Y gastric bypass. Surg Endosc. 2012 Jul;26(7):1997-2002. doi: 10.1007/s00464-011-2140-0. Epub 2012 Jan 19. PMID 22258299
- [Background] Kellogg TA. Revisional bariatric surgery. Surg Clin North Am. 2011 Dec;91(6):1353-71, x. doi: 10.1016/j.suc.2011.08.004. PMID 22054158
- [Background] deWolfe MA, Bower CE. Using the StomaphyX(TM) endoplicator to treat a gastric bypass complication. JSLS. 2011 Jan-Mar;15(1):109-13. doi: 10.4293/108680811X13022985131570. PMID 21902955
- [Background] Thompson CC, Jacobsen GR, Schroder GL, Horgan S. Stoma size critical to 12-month outcomes in endoscopic suturing for gastric bypass repair. Surg Obes Relat Dis. 2012 May-Jun;8(3):282-7. doi: 10.1016/j.soard.2011.03.014. Epub 2011 Apr 19. PMID 21640665
- [Background] Raman SR, Holover S, Garber S. Endolumenal revision obesity surgery results in weight loss and closure of gastric-gastric fistula. Surg Obes Relat Dis. 2011 May-Jun;7(3):304-8. doi: 10.1016/j.soard.2011.01.045. Epub 2011 Feb 22. PMID 21474389
- [Background] Heneghan HM, Yimcharoen P, Brethauer SA, Kroh M, Chand B. Influence of pouch and stoma size on weight loss after gastric bypass. Surg Obes Relat Dis. 2012 Jul-Aug;8(4):408-15. doi: 10.1016/j.soard.2011.09.010. Epub 2011 Sep 23. PMID 22055390
- [Background] Yimcharoen P, Heneghan HM, Singh M, Brethauer S, Schauer P, Rogula T, Kroh M, Chand B. Endoscopic findings and outcomes of revisional procedures for patients with weight recidivism after gastric bypass. Surg Endosc. 2011 Oct;25(10):3345-52. doi: 10.1007/s00464-011-1723-0. Epub 2011 Apr 30. PMID 21533520

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 patients were recruited 23 underwent the proposed procedure
Groups:
- All Study Participants: Patients who previously underwent bariatric surgery who failed to lose the expected weight or regained weight.
  Endoscopic Suturing to Create Early Satiety: Evaluating the efficacy of endoscopic suturing for weight loss.
Period: Overall Study
Arm/Group | All Study Participants
Started | 24
Underwent Procedure | 23
Completed | 23
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Weight Gain
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 47.6 [33 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Weight Loss
Description: We will track patient's weight after their endoscopic bariatric surgery.
Time Frame: 3 months after procedure
Measure: Mean (Full Range); unit: Pounds
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Pounds | 13.3 [0 to 40]

2. Secondary Outcome: Number of Participants With Resolved Co-morbidities
Description: We will track the patient's weight loss and see if their obesity-related co-morbidities resolve.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Patients who previously underwent bariatric surgery who failed to lose the expected weight or regained weight.
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Participants | 23

3. Secondary Outcome: Tolerance
Description: We will be monitoring patient's tolerance to this procedure and evaluate their satisfaction via a short questionnaire.
Time Frame: 2 years
Population: Data were not collected for this outcome measure. Milestone visit dates at which surveys were going to be provided were not followed through by patients resulting in the lack of data collected.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Weight Gain
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weight Gain (N=24)
Leak (Gastrointestinal disorders) | 1 — The patient sustained a small leak from the revision. This was identified the day after surgery and treated with IV antibiotics. She recovered 4 days afterwards and was discharged. We followed her for 3 hours and she has been doing well.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Gain (N=24)
Dysphagia (Gastrointestinal disorders) | 1 (1) — Patient's revision was very tight. We dilated her and it resolved. No long term issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT01871896/Prot_SAP_000.pdf